CLINICAL TRIAL: NCT03061240
Title: Smart Pain Assesment Tool Based on Internet of Things
Acronym: SPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turku (Other)
Collaborators: Academy of Finland (Other); Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Sanna Salanterä, Professor, University of Turku
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 29092016
Record Dates: First submitted 2017-02-09; First posted 2017-02-23 (Actual); Last update posted 2018-12-24 (Actual); Status verified 2018-12

CONDITIONS: Pain
Keywords: Internet of Things
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Postoperative patients (Experimental): We recruit postoperative patients who undergo open surgery and are not receiving local anesthesia. We install a smart pain assessment tool on patient's skin to capture different type of data.
  Interventions: Device: Smart pain assessment tool

INTERVENTIONS:
Device: Smart pain assessment tool — We record and analyze multiple bio-signals from post-operative patients in the attempt to evaluate their experienced pain.

SUMMARY:
This study is the second phase of a research project called "Smart Pain Assessment Tool based on Internet-of-Things". During the course of this project, a smart pain assessment tool (SPA) to detect and assess pain employing behavioural and physiologic indicators will be developed. We aim to assess pain based on changes in electromyographic (EMG) activity in facial muscles, i.e. changes in facial expressions and simultaneously use physiologic signs such as heart rate, respiratory rate and galvanic skin response as adjuvant measures to develop an algorithm for pain assessment in critically ill patients.

DETAILED DESCRIPTION:
The aim of this "smart pain assessment tool based on internet of things" SPA-research project is to develop an automatic and versatile pain assessment tool algorithm for detection and assessment of pain in a reliable and objective way in non-communicative patients. The final objective of the research project is to develop a smart pain assessment tool to detect and assess pain employing behavioural and physiologic indicators for a wide range of users/patients from infants to elderly people who are unable to communicate normally. The research project consists of three clinical phases (European Commision. Meddev 2.7/4/2010). The clinical phase I of the research project focused on developing pain assessment techniques involuntary working-age healthy study subjects. This current Clinical phase II includes the further development and research of the smart pain assessment tool in elective (non emergency) postoperative surgical patients during their stay after surgery in a recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Subject is scheduled for major surgery that requires general anesthesia and is likely to cause moderate to severe pain postoperatively which needs to be treated with systemic analgesics
* Ability to communicate
* Written informed consent
* Healthy facial skin

Exclusion Criteria:

* Subject treated with local anesthesia during surgery
* Any diagnosed condition affecting cognitive functions
* Surgery affecting hands where pulse oximetry and galvanic skin reaction are recorded or areas where facial muscle activity is measured
* Any diagnosed condition affecting central nervous system, facial nerves or muscles.
* Significant facial hair growth in the area where the sensors will be attached
* Tattoos in the area where the sensors will be attached

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2017-11-20 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Facial muscle activity | 2 hours after surgery when the subject has woken up
  The device is designed for multi-channel EMG acquisition from facial skin. Measuring a combination of EMG signals and their energy level (amplitude).

SECONDARY OUTCOMES:
Skin conductance | 2 hours after surgery when the subject has woken up
  Galvanic skin response (GSR), also known as electrodermal activity (EDA) or skin conductance (SC).
Pain assesment by VAS | 2 hours after surgery when the subject has woken up
  Subjective feeling of pain is asked every 10 minutes by using numeric visual analog scale (VAS), values are given from 0-10.
Heart rate | 2 hours after surgery when the subject has woken up
  Heart rate is monitored and recorded.
Respiratory rate | 2 hours after surgery when the subject has woken up
  Respiratory rate is monitored and recorded.
Oxygen saturation | 2 hours after surgery when the subject has woken up
  Oxygen saturation is monitored and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Salanterä, Prof, Principal Investigator — University of Turku
Locations (1):
- University of Turku, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jeitziner MM, Schwendimann R, Hamers JP, Rohrer O, Hantikainen V, Jakob SM. Assessment of pain in sedated and mechanically ventilated patients: an observational study. Acta Anaesthesiol Scand. 2012 May;56(5):645-54. doi: 10.1111/j.1399-6576.2012.02660.x. Epub 2012 Mar 7. PMID 22404146
- [Background] Viertio-Oja H, Maja V, Sarkela M, Talja P, Tenkanen N, Tolvanen-Laakso H, Paloheimo M, Vakkuri A, Yli-Hankala A, Merilainen P. Description of the Entropy algorithm as applied in the Datex-Ohmeda S/5 Entropy Module. Acta Anaesthesiol Scand. 2004 Feb;48(2):154-61. doi: 10.1111/j.0001-5172.2004.00322.x. No abstract available. PMID 14995936
- [Background] Prkachin KM. Assessing pain by facial expression: facial expression as nexus. Pain Res Manag. 2009 Jan-Feb;14(1):53-8. doi: 10.1155/2009/542964. PMID 19262917
- [Background] Ledowski T, Ang B, Schmarbeck T, Rhodes J. Monitoring of sympathetic tone to assess postoperative pain: skin conductance vs surgical stress index. Anaesthesia. 2009 Jul;64(7):727-31. doi: 10.1111/j.1365-2044.2008.05834.x. Epub 2009 Jan 28. PMID 19183409
- [Background] EPoSS. 2008. Internet of Things in 2020: a Roadmap for the Future. European Technology Platform on Smart Systems Integration. European Commission Information Society.